CLINICAL TRIAL: NCT02095665
Title: Ureteral Stent-related Pain and Mirabegron (SPAM) Trial
Acronym: SPAM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPAM
Record Dates: First submitted 2014-02-17; First posted 2014-03-26 (Estimated); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Nephrolithiasis
Keywords: ureteric stents; LUTS; lower urinary tract symptoms
MeSH Terms: conditions — Nephrolithiasis; Lower Urinary Tract Symptoms | interventions — mirabegron; Tamsulosin; Acetaminophen

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Narcotic analegesic only (Active Comparator): Drug:
  Tylenol #3 1 tablet every six hours as necessary
  Interventions: Drug: Tylenol #3
- Mirabegron and narcotic analgesia (Active Comparator): Drug :
  Mirabegron 50 mg oral daily
  Drug:
  Tylenol #3 1 tablet every six hours as necessary
  Interventions: Drug: Mirabegron; Drug: Tylenol #3
- Tamsulosin and narcotic analgesia (Active Comparator): Drug:
  Tamsulosin 0.4mg oral daily Drug: Tylenol #3 1 tablet every six hours as necessary
  Interventions: Drug: Tamsulosin; Drug: Tylenol #3
- Mirabegron, Tamsulosin and narcotic (Experimental): Drug:
  Mirabegron 50 mg oral daily
  Drug:
  Tamsulosin 0.4mg oral daily
  Drug:
  Tylenol #3 1 tablet every six hours as necessary
  Interventions: Drug: Mirabegron; Drug: Tamsulosin; Drug: Tylenol #3

INTERVENTIONS:
Drug: Mirabegron — 50 mg of Mirabegron daily from stent insertion until removal 5 to 10 days
  Other Names: Myrbertiq
  Arms: Mirabegron and narcotic analgesia; Mirabegron, Tamsulosin and narcotic
Drug: Tamsulosin — 0.4 mg of Tamsulosin daily and 1 tab of Percocet every 4 hours as necessary from stent insertion until removal 5 to 10 days
  Other Names: Flomax
  Arms: Mirabegron, Tamsulosin and narcotic; Tamsulosin and narcotic analgesia
Drug: Tylenol #3 — 1 tab of Tylenol #3 every 6 hours as necessary from stent insertion until removal 5 to 10 days
  Other Names: Atasol

SUMMARY:
Ureteric stents are used often following ureteroscopy for prevention of obstruction from edema and or stone fragments. They are often associated with pain, voiding often, the need to urinate quickly and finding blood in the urine called "lower urinary tract symptoms" or LUTS for short. There is randomized studies showing the efficacy of α-blockers such as tamsulosin in relieving "stent symptoms" (pain and LUTS). There is emerging but limited evidence to show that antimuscarinic medications, used to treat overactive bladder (OAB) have some efficacy in decreasing stent symptoms. Mirabegron is a beta-agonist used to decrease OAB symptoms.

Mirabegron functions to mediate relaxation of the detrusor muscle and has been useful in treating OAB symptoms. Conventional antimuscarinic medications often have bothersome side effects like dry mouth, constipation, blurred vision and cognitive impairment. This may limit their use in some populations. Mirabegron is well-tolerated with a good safety profile and therefore may be useful in treating stent symptoms without the bothersome side effects commonly seen with antimuscarinic medications. .

The investigators hypothesize that mirabegron is effective in decreasing ureteral stent related LUTS and pain.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* First presentation for ureteroscopy for this particular stone
* Planned insertion of double J ureteral stent
* Planned ureteral stenting ≥5 days
* Follow-up conducted at the Queen Elizabeth II Health Sciences Centre

Exclusion Criteria:

* Bilateral ureteral stents to be inserted
* Stent already in situ prior to ureteroscopy
* Patients with congenital renal abnormalities (ie: horseshoe kidney, ectopic kidney, etc)
* Patients with urinary diversion
* Patients with a history of interstitial cystitis/painful bladder syndrome, chronic prostatitis, or neurogenic bladder
* Indwelling foley catheter
* Active urinary tract infection
* Patients currently taking antimuscarinics, mirabegron, or α-blockers
* Patients with contraindications to receiving either mirabegron or tamsulosin (ie: urinary retention, end-stage renal disease, orthostatic hypotension, uncontrolled hypertension, known QT prolongation, severe aortic regurgitation), significant cognitive impairment, pregnancy, and active urinary tract infection
* Planned upcoming elective cataract surgery
* Suspected or confirmed ureteral perforation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2018-03-23 (Actual); Study Completion 2018-03-23 (Actual)

PRIMARY OUTCOMES:
Ureteral stent related pain and lower urinary tract symptoms (LUTS) as measured by the Ureteral Stent Symptom Questionnaire. | Measured twice, once at the time of surgery when stent is inserted and secondly at the time the stent is removed which will occur 5 to 10 days following surgery.
  The primary objective of this study is to determine if mirabegron is effective in decreasing ureteral stent related lower urinary tract symptoms (LUTS) following ureteroscopy for urolithiasis when compared to tamsulosin alone and in combination. Utilizing the Ureteral Stent Symptom Questionnaire, a self-administered questionnaire participants will report their urinary symptoms for comparison, enabling the comparison through out the different treatment arms.

SECONDARY OUTCOMES:
Quality of life impact of mirabegron for stent symptoms as measured with the Ureteral Stent Symptoms Questionnaire. | Measured twice, once at the time of surgery when stent is inserted and secondly at the time the stent is removed occuring 5 to 10 days later.
  The secondary objectives are to determine if mirabegron is effective in decreasing ureteral stent related pain compared to tamsulosin alone and in combination following ureteroscopy for urolithiasis, determining if there are any improvements in health related quality of life (HRQoL). Subjects will maintain a diary recording the frequency of pain medication through out the period the stent remains insitu, 5 to 10 days.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea G Lantz, MD, Principal Investigator — Staff Urologist
Locations (1):
- Nova Scotia Health Authority, Central, Halifax, Nova Scotia, Canada